CLINICAL TRIAL: NCT06371404
Title: Imaging Traumatic Stress and Alcohol Use Disorder With [18F]Bavarostat
Status: Recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2000037129; 1U54AA027989-01 (NIH)
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Alcohol Use Disorder; Post Traumatic Stress Disorder
MeSH Terms: conditions — Alcoholism; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (5):
- PTSD: Subjects with Post Traumatic Stress Disorder
  Interventions: Drug: Bavarostat
- AUD: Subjects with Alcohol Use Disorder
  Interventions: Drug: Bavarostat
- PTSD & AUD: Subjects with Post Traumatic Stress Disorder and Alcohol Use Disorder
  Interventions: Drug: Bavarostat
- HC: Healthy Control Subjects
  Interventions: Drug: Bavarostat
- TC: Trauma-exposed healthy control subjects.
  Interventions: Drug: Bavarostat

INTERVENTIONS:
Drug: Bavarostat — Up to two injections of ≤ 5 mCi [F18] Bavarostat

SUMMARY:
The overall objective of this study it to use Positron Emission Tomography (PET) brain imaging and a radiotracer that measures the epigenetic marker Histone Deacetylase 6 (HDAC6) to examine HDAC6 expression in people with Post-Traumatic Stress Disorder (PTSD), Alcohol Use Disorder (AUD), or concurrent PTSD and AUD with control groups. While there are a large number of studies conducted in preclinical stress and addiction models, these findings have not been translated to people living with these disorders. This study will examine relationships between HDAC6 and clinical variables of interest. Findings could direct treatment development.

DETAILED DESCRIPTION:
This study will image 150 subjects total, as outlined below. Subjects will be asked to participate in magnetic resonance imaging (MRI) and PET imaging procedures as well as behavioral and cognitive tasks to better understand stress and alcohol related behaviors. MRI is required to detect significant brain abnormalities and for use in the PET image analysis.

In Aim 1, Up to 30 PTSD and 30 TC will be imaged with [18F]Bavarostat to measure levels of HDAC6 throughout the brain to determine whether individuals with PTSD have altered levels of HDAC6 expression compared to trauma-exposed healthy controls.

In Aim 2, Up to 30 AUD and 30 HC will be imaged with [18F]Bavarostat to measure levels of HDAC6 throughout the brain to determine whether individuals with AUD have altered levels of HDAC6 expression compared to healthy controls.

In Aim 3, Up to 30 comorbid PTSD & AUD subjects will be imaged with [18F]Bavarostat to measure levels of HDAC6 throughout the brain to determine whether individuals with comorbid PTSD & AUD have altered levels of HDAC6 expression compared to trauma-exposed healthy controls.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give voluntary written informed consent
2. Is able to read and write, able to communicate effectively with the investigator, and comply with all study requirements, restrictions, and directions of the research staff
3. Men or women, aged 18 to 70, at screening
4. In good general health as evidenced by medical history, physical examination, ECG, serum/urine biochemistry, hematology, and serology tests
5. Participants with PTSD will have a current diagnosis of PTSD according to DSM-5 criteria (CAPS-5 ascertained diagnosis, confirmed by the Principal Investigators. TC subjects must have a DSM-5 criteria traumatic event with no PTSD diagnosis
6. Participants with AUD will have a current diagnosis of AUD according to DSM-5 criteria (i.e., SCID-5 ascertained diagnosis, confirmed by the Principal Investigators);
7. Participants with AUD will meet the following drinking criteria: males will drink > 14 drinks per week and exceed 4 drinks per day at least twice per week; females will drink > 7 drinks per week and exceed 3 drinks per day at least twice per week. They must meet drinking criteria during a consecutive 30-day period within the 90 days prior to intake.
8. Healthy subjects will have no current or past diagnosis of AUD or other significant substance use disorder. They will drink less than 5 alcoholic drinks per week with no heavy drinking days (i.e., >4 drinks/day for men; >3 drinks/day for women) in the last 30 days;

Exclusion Criteria:

1. Current significant medical condition such as neurological, cardiovascular, endocrine, renal, liver, or thyroid pathology that would impact the integrity of the data (note that elevated liver enzymes for individuals with AUD will not be exclusionary)
2. Past or current neurological disorder or disorders affecting the brain including but not limited to multiple sclerosis, history of stroke, brain tumors, traumatic brain injury with loss of consciousness, seizure disorder;
3. Current significant psychiatric disorder including severe substance use disorder (other than alcohol or tobacco use disorders*), and past or current psychotic symptoms,
4. Regular use in the past 6 months of any prescription, psychoactive or herbal medications (e.g., antidepressants, antipsychotics, anxiolytics) that would impact the integrity of the data (e.g., naltrexone); No subject will be asked to stop taking medication to participate in the study;
5. Pregnancy or lactation
6. Blood donation within eight weeks of the start of the study.
7. History of a bleeding disorder or are currently taking anticoagulants (such as Coumadin, Heparin, Pradaxa, Xarelto).
8. Unable to safely discontinue or hold aspirin and other NSAID use
9. MRI incompatible implants (i.e., such as pacemaker, artificial joints, non-removable body piercings) and other contraindications for MRI, such as claustrophobia, having implanted or embedded metal objects/fragments or fragments in the head or body that would present a risk during the MRI scanning procedure, or have worked with ferrous metals either as a vocation or hobby (for example, as a sheet metal worker, welder, or machinist).
10. Participation in other research studies involving inonizing radiation within one year of the PET scans that would cause the subject to exceed the yearly dose limits for healthy volunteers.
11. Subject who has current, past, or anticipated exposure to radiation in the work place within one year of the proposed research scans that in combination with the study tracer would result in a cumulative exposure that exceeds recommended exposure limits.
12. Has any condition that, in the opinion of the investigator, would prevent compliance with the study protocol.
13. History of complicated alcohol withdrawal including history of delirium tremens; seizure, hospitalization for withdrawal.
14. Alcohol intoxication at time of screening.
15. A CIWA score ≥8 at intake or on scan day.
16. Subjects who are, in the opinion of the study physician, unable to safely abstain from alcohol overnight prior to their study visits.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 150 adult male and female subjects, aged 18-70, who are in general good health, meet the inclusion criteria, and who do not meet any of the exclusion criteria will be eligible for enrollment into Aim 1, Aim 2, or Aim 3 of the study.
  Up to 30 PTSD and 30 TC subjects will be enrolled into Aim 1 of the study. Up to 30 AUD and 30 HC subjects will be enrolled into Aim 2 of the study. Up to 30 comorbid PTSD & AUD subjectswill be enrolled into Aim 3 of the study.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2030-06-01 (Estimated); Study Completion 2031-06-01 (Estimated)

PRIMARY OUTCOMES:
HDAC6 expression in people with Post-Traumatic Stress Disorder | Baseline
HDAC6 expression in people with Alcohol use Disorder | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided